CLINICAL TRIAL: NCT02632708
Title: A Phase 1, Multicenter, Open-Label, Safety Study of AG-120 or AG-221 in Combination With Induction Therapy and Consolidation Therapy in Patients With Newly Diagnosed Acute Myeloid Leukemia With an IDH1 and/or IDH2 Mutation
Brief Title: Safety Study of AG-120 or AG-221 in Combination With Induction and Consolidation Therapy in Participants With Newly Diagnosed Acute Myeloid Leukemia (AML) With an IDH1 and/or IDH2 Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG120-221-C-001; 2015-004290-33 (EudraCT Number)
Record Dates: First submitted 2015-11-19; First posted 2015-12-17 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Newly Diagnosed Acute Myeloid Leukemia (AML); Untreated AML; AML Arising From Myelodysplastic Syndrome (MDS); AML Arising From Antecedent Hematologic Disorder (AHD); AML Arising After Exposure to Genotoxic Injury
Keywords: Acute Myeloid Leukemia; AML; Untreated AML; De novo AML; Secondary AML; Newly diagnosed AML; IDH1; IDH2; Induction therapy; Consolidation therapy; IDH
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib; enasidenib; Cytarabine; Daunorubicin; Idarubicin; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- AG-120 with cytarabine and daunorubicin (Experimental): Daily AG-120 administered orally in combination with standard Induction therapy and consolidation therapy. After 1 cycle of induction therapy, participants may undergo a second induction cycle given as per institutional practice. Participants who achieve an adequate response at the end of induction therapy will go on to receive consolidation therapy (mitoxantrone/etoposide or up to 4 cycles of cytarabine) in combination with AG-120. Participants who complete consolidation therapy and are in complete response (CR) or complete remission with incomplete hematologic recovery (CRi) (including CR with incomplete platelet recovery [CRp]) may continue on maintenance therapy and receive daily treatment with AG-120.
  Interventions: Drug: AG-120; Drug: cytarabine; Drug: daunorubicin; Drug: mitoxantrone; Drug: etoposide
- AG-120 with cytarabine and idarubicin (Experimental): Daily AG-120 administered orally in combination with standard Induction therapy and consolidation therapy. After 1 cycle of induction therapy, participants may undergo a second induction cycle given as per institutional practice. Participants who achieve an adequate response at the end of induction therapy will go on to receive consolidation therapy (mitoxantrone/etoposide or up to 4 cycles of cytarabine) in combination with AG-120. Participants who complete consolidation therapy and are in CR or CRi (including CRp) may continue on maintenance therapy and receive daily treatment with AG-120.
  Interventions: Drug: AG-120; Drug: cytarabine; Drug: idarubicin; Drug: mitoxantrone; Drug: etoposide
- AG-221 with cytarabine and daunorubicin (Experimental): Daily AG-221 administered orally in combination with standard Induction therapy and consolidation therapy. After 1 cycle of induction therapy, participants may undergo a second induction cycle given as per institutional practice. Participants who achieve an adequate response at the end of induction therapy will go on to receive consolidation therapy (mitoxantrone/etoposide or up to 4 cycles of cytarabine) in combination with AG-221. Participants who complete consolidation therapy and are in CR or CRi (including CRp) may continue on maintenance therapy and receive daily treatment with AG-221.
  Interventions: Drug: AG-221; Drug: cytarabine; Drug: daunorubicin; Drug: mitoxantrone; Drug: etoposide
- AG-221 with cytarabine and idarubicin (Experimental): Daily AG-221 administered orally in combination with standard Induction therapy and consolidation therapy. After 1 cycle of induction therapy, participants may undergo a second induction cycle given as per institutional practice. Participants who achieve an adequate response at the end of induction therapy will go on to receive consolidation therapy (mitoxantrone/etoposide or up to 4 cycles of cytarabine) in combination with AG-221. Participants who complete consolidation therapy and are in CR or CRi (including CRp) may continue on maintenance therapy and receive daily treatment with AG-221.
  Interventions: Drug: AG-221; Drug: cytarabine; Drug: idarubicin; Drug: mitoxantrone; Drug: etoposide
- AG-221 (starting on Day 8) with cytarabine and daunorubicin (Experimental): Daily AG-221 administered orally starting on Day 8 of induction cycle 1 in combination with standard Induction therapy and consolidation therapy. After 1 cycle of induction therapy, participants may undergo a second induction cycle given as per institutional practice. Participants who achieve an adequate response at the end of induction therapy will go on to receive consolidation therapy (mitoxantrone/etoposide or up to 4 cycles of cytarabine) in combination with AG-221. Participants who complete consolidation therapy and are in CR or CRi (including CRp) may continue on maintenance therapy and receive daily treatment with AG-221.
  Interventions: Drug: AG-221; Drug: cytarabine; Drug: daunorubicin; Drug: mitoxantrone; Drug: etoposide
- AG-221 (starting on Day 8) with cytarabine and idarubicin (Experimental): Daily AG-221 administered orally starting on Day 8 of induction cycle 1 in combination with standard Induction therapy and consolidation therapy. After 1 cycle of induction therapy, participants may undergo a second induction cycle given as per institutional practice. Participants who achieve an adequate response at the end of induction therapy will go on to receive consolidation therapy (mitoxantrone/etoposide or up to 4 cycles of cytarabine) in combination with AG-221. Participants who complete consolidation therapy and are in CR or CRi (including CRp) may continue on maintenance therapy and receive daily treatment with AG-221.
  Interventions: Drug: AG-221; Drug: cytarabine; Drug: idarubicin; Drug: mitoxantrone; Drug: etoposide

INTERVENTIONS:
Drug: AG-120
  Arms: AG-120 with cytarabine and daunorubicin; AG-120 with cytarabine and idarubicin
Drug: AG-221
  Arms: AG-221 (starting on Day 8) with cytarabine and daunorubicin; AG-221 (starting on Day 8) with cytarabine and idarubicin; AG-221 with cytarabine and daunorubicin; AG-221 with cytarabine and idarubicin
Drug: cytarabine
Drug: daunorubicin
  Arms: AG-120 with cytarabine and daunorubicin; AG-221 (starting on Day 8) with cytarabine and daunorubicin; AG-221 with cytarabine and daunorubicin
Drug: idarubicin
  Arms: AG-120 with cytarabine and idarubicin; AG-221 (starting on Day 8) with cytarabine and idarubicin; AG-221 with cytarabine and idarubicin
Drug: mitoxantrone
Drug: etoposide

SUMMARY:
The purpose of this Phase I, multicenter, clinical trial is to evaluate the safety of AG-120 and AG-221 when given in combination with standard AML induction and consolidation therapy. The study plans to evaluate up to 2 dose levels of AG-120 in participants with an isocitrate dehydrogenase protein 1 (IDH1) mutation and up to 2 dose levels of AG-221 in participants with an isocitrate dehydrogenase protein 2 (IDH2) mutation. AG-120 or AG-221 will be administered with 2 types of AML induction therapies (cytarabine with either daunorubicin or idarubicin) and 2 types of AML consolidation therapies (mitoxantrone with etoposide [ME] or cytarabine). After consolidation therapy, participants may continue on to maintenance therapy and receive daily treatment with single-agent AG-120 or AG-221 until relapse, development of an unacceptable toxicity, or hematopoietic stem cell transplant (HSCT). The study will end when all participants have discontinued study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must ≥18 years of age
* Previously untreated AML (de novo or secondary) defined according to World Health Organization (WHO) criteria, excluding acute promyelocytic leukemia (APL) [AML with t(15;17)], with locally documented IDH1 and/or IDH2 gene mutation scheduled for induction therapy followed by consolidation therapy. Participants with secondary AML is defined as AML arising after myelodysplastic syndromes (MDSs) or other antecedent hematologic disorders (AHDs) or AML arising after exposure to genotoxic injury including radiation and/or chemotherapy are also eligible. Participants may have had previous treatment for MDS or other AHD, including hypomethylating agents (HMAs), provided it was ≥ 14 days prior to study drug initiation
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 2
* Adequate hepatic function as evidenced by: serum total bilirubin ≤1.5 × upper limit of normal (ULN) unless considered due to Gilbert's disease, a gene mutation in UGT1A1 (only for patients who will be receiving AG-221), or leukemic involvement following approval by the study Sponsor; aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3.0 × ULN, unless considered due to leukemic involvement following approval by the study Sponsor
* Adequate renal function as evidenced by serum creatinine ≤2.0 × ULN or creatinine clearance 40 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR)
* Agree to serial blood and bone marrow sampling
* Meet any criteria necessary for the safe and proper use of the induction and consolidation agents involved in this trial
* Able to understand and willing to sign an informed consent form. A legally authorized representative may consent on behalf of a participant who is otherwise unable to provide informed consent, if acceptable to, and approved by, the site's Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Female participants with reproductive potential must agree to undergo a medically supervised pregnancy test prior to starting study drug. The first pregnancy test will be performed at screening (within 7 days prior to first study drug administration). A pregnancy test should also be performed on the day of the first study drug administration and confirmed negative prior to dosing as well as before dosing on Day 1 of all subsequent cycles
* Female participants with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of the therapy. Participants with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal for at least 24 consecutive months. Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use one highly effective form (for participants receiving AG-221) or two highly effective forms (for participants receiving AG-120) of contraception from the time of giving informed consent, during the study, and for 2 months (for participants receiving AG-221) and for 4 months (for participants receiving AG-120) following the last dose of AG-120 or AG-221 (females and males). A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier method (e.g., synthetic condoms, diaphragm or cervical cap with spermicidal foam, cream, or gel) or male partner sterilization

Exclusion Criteria:

* Prior chemotherapy for AML. Hydroxyurea is allowed prior to enrollment for the control of peripheral leukemic blasts in participants with leukocytosis; hydroxyurea may be allowed on study with study Sponsor approval
* Taking medications with narrow therapeutic windows, unless they can be transferred to other medications prior to enrolling or unless the medications can be properly monitored during the study
* Taking known strong cytochrome P450 (CYP) 3A4 inducers, unless they can be transferred to other medications prior to enrolling. For participants taking AG-120, systemic administration of a moderate or strong CYP3A4 inhibitor requires careful monitoring of the heart rate-corrected QT interval (QTc) using Fridericia's formula (QTcF)
* Taking P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) or OATP1B1/1B3 transporter-sensitive substrate medications unless they can be transferred to alternative medications within ≥5 half-lives prior to administration of AG-221, or unless the medications can be adequately monitored during the study. There are no restrictions regarding the co-administration of such medications with AG-120.
* Pregnant or breastfeeding
* Uncontrolled active infection or uncontrolled invasive fungal infection (positive blood or tissue culture). An infection controlled with an approved or closely monitored antibiotic/antifungal treatment is allowed
* Prior history of malignancy, other than MDS or AML, unless the participant has been free of the disease for ≥1 year prior to the start of study treatment However, participants with the following history/concurrent conditions are allowed: basal or squamous cell carcinoma of the skin; carcinoma in situ of the cervix; carcinoma in situ of the breast; incidental histologic finding of prostate cancer
* Significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) Class III or IV congestive heart failure; myocardial infarction, unstable angina and/or stroke; or left ventricular ejection fraction (LVEF) <40% by echocardiogram (ECHO), or by other methods according to institutional practice, obtained within 28 days prior to the start of study treatment
* QTc interval using Fridericia's formula (QTcF) ≥450 milliseconds (msec) or other factors that increase the risk of QT interval prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Bundle branch block and prolonged QTc are permitted with approval of the study Sponsor
* Taking medications that are known to prolong the QT interval unless they can be transferred to other medications within ≥5 half-lives prior to dosing (If equivalent medication is not available QTc will be closely monitored)
* Known infection caused by human immunodeficiency virus (HIV) or active hepatitis B or C
* Dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs
* Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid (CSF) during screening is required only if there is a clinical suspicion of CNS involvement by leukemia during screening.
* Immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Any other medical or psychological condition deemed by the Investigator to be likely to interfere with a participant's ability to give informed consent or participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 26 weeks
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of AG-120 and AG-221 when Administered with Induction and Consolidation Therapy | Up to 26 weeks
Pharmacokinetics (PK) of AG-120 and AG-221 in Plasma when Administered with Induction and Consolidation Therapy | Up to 26 weeks
  Descriptive statistics will be used to summarize PK parameters for each dose group and, where appropriate, for the entire population.
2-hydroxyglutarate (2-HG) Levels in Plasma | Up to 26 weeks
Clinical Activity of AG-120 and AG-221 According to the 2003 Revised International Working Group (IWG) Criteria for AML | Up to 26 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- United States (14):
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Universitatsklinikum Ulm, Ulm, Germany
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Stein EM, DiNardo CD, Fathi AT, Mims AS, Pratz KW, Savona MR, Stein AS, Stone RM, Winer ES, Seet CS, Dohner H, Pollyea DA, McCloskey JK, Odenike O, Lowenberg B, Ossenkoppele GJ, Patel PA, Roshal M, Frattini MG, Lersch F, Franovic A, Nabhan S, Fan B, Choe S, Wang H, Wu B, Hua L, Almon C, Cooper M, Kantarjian HM, Tallman MS. Ivosidenib or enasidenib combined with intensive chemotherapy in patients with newly diagnosed AML: a phase 1 study. Blood. 2021 Apr 1;137(13):1792-1803. doi: 10.1182/blood.2020007233. PMID 33024987
- [Derived] Montesinos P, Fathi AT, de Botton S, Stein EM, Zeidan AM, Zhu Y, Prebet T, Vigil CE, Bluemmert I, Yu X, DiNardo CD. Differentiation syndrome associated with treatment with IDH2 inhibitor enasidenib: pooled analysis from clinical trials. Blood Adv. 2024 May 28;8(10):2509-2519. doi: 10.1182/bloodadvances.2023011914. PMID 38507688
- [Derived] Fan B, Chen Y, Yin F, Hua L, Almon C, Nabhan S, Cooper M, Yang H, Hossain M. Pharmacokinetic/Pharmacodynamic Evaluation of Ivosidenib or Enasidenib Combined With Intensive Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed IDH1/2-Mutant Acute Myeloid Leukemia. Clin Pharmacol Drug Dev. 2022 Apr;11(4):429-441. doi: 10.1002/cpdd.1067. Epub 2022 Feb 14. PMID 35166065
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/